CLINICAL TRIAL: NCT00968084
Title: Screening Protocol for Subjects Being Evaluated for Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) Protocols
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090201; 09-H-0201
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10-25

CONDITIONS: Inflammatory Disease; Autoimmune Disease; Immunologic Disease; Healthy Volunteers
Keywords: Diagnostic Work Up; Normal Volunteers; HV; Inflammatory Disease; Autoimmune Disease; Immunologic Disease; Healthy Volunteer
MeSH Terms: conditions — Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* For every CHI research study, patients must fulfill a list of criteria, based primarily on their medical condition. To determine whether a patient meets these eligibility criteria to participate in a research protocol, researchers must perform a series of diagnostic tests and procedures.
* These evaluations are designed to evaluate a participant s general medical condition (i.e., blood tests, function of certain organs such as the lungs, heart, liver, or kidneys), and to confirm a diagnosis or ensure that a healthy volunteer is in good condition. They maximize the safety for the patients and healthy volunteers at CHI.

Objective:

- To determine the eligibility of patients and healthy volunteers for active CHI research protocols.

Eligibility:

* The procedures included in this protocol will determine eligibility for active CHI research protocols.
* Both healthy volunteers and patients will be evaluated.

Design:

* Required tests and procedures for various research studies may include the following: history and physical examination, blood and urine tests, lung and heart function tests (echocardiogram, electrocardiogram, stress test), imaging studies (X-rays, magnetic resonance imaging (MRI), computerized tomography (CT), and tissue collection.
* Participants will be asked to undergo tests only for the study or studies for which they are being considered. The research team will provide further information on any additional tests that may be required.
* After all eligibility assessments are complete, participants may be offered participation in one or more CHI research protocols or referred back to a home physician.

DETAILED DESCRIPTION:
This protocol is designed for screening of subjects prior to a decision as to their eligibility for participation on a Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) tissue procurement or investigative therapy protocol. The purpose of the protocol is to allow investigation into any underlying immunologic and/or inflammatory processes and to assess the status of organ systems, important both to determine suitability for participation on specific protocols and/or ability to safely tolerate tissue procurement or investigative treatments and procedures. It also allows the investigation as to whether subjects are eligible for participation as a volunteer based on eligibility criteria that include generally good health status by history and physical examination and laboratory assessment. After completion of the screening process, the subject will either be offered an opportunity to participate in a specific research protocol, or if no appropriate protocol is identified, will have recommendations for other treatment options conveyed to the primary or referring physician.

Primary objective is to determine subject eligibility for participation on Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) tissue procurement or investigative therapy protocols.

Primary endpoint is the results of clinical, imaging and laboratory assessments.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosed with a disorder for which the CHI has an active research protocol, and based on information received from an outside physician, the patient appears to meet at least preliminary eligibility criteria for that protocol.

     OR

     Self proclaimed healthy volunteer for whom the CHI has a study actively recruiting healthy volunteers and he/she appears to meet preliminary eligibility as a healthy volunteer.
  2. Age greater than or equal to 2 (healthy volunteers greater than or equal to 8)
  3. Weight greater than 12 kg
  4. The subject or the subject s guardian is capable of informed consent, and willing to sign the consent form after initial counseling by clinical staff. Separate consent forms for all interventional or surgical procedures will be obtained after explanation of the specific procedure.

EXCLUSION CRITERIA:

All subjects not fulfilling the inclusion criteria will be considered ineligible.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2009-08-06; Study Completion 2017-10-25

PRIMARY OUTCOMES:
Results of clinical, imaging and laboratory assessments.

SECONDARY OUTCOMES:
Eligibility for participation on Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) tissue procurement of investigative therapy protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] El-Chemaly S, Cheung F, Kotliarov Y, O'Brien KJ, Gahl WA, Chen J, Perl SY, Biancotto A, Gochuico BR. The Immunome in Two Inherited Forms of Pulmonary Fibrosis. Front Immunol. 2018 Jan 31;9:76. doi: 10.3389/fimmu.2018.00076. eCollection 2018. PMID 29445374